CLINICAL TRIAL: NCT02549937
Title: A Multi-Center, Open-Label, Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of Surufatinib (HMPL-012), Previously Named Sulfatinib in Advanced Solid Tumors
Brief Title: A Multi-Center, Open-Label Study of Surufatinib (HMPL-012) in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2015-012-00US1
Expanded Access: NCT04814732 (No longer available)
Record Dates: First submitted 2015-07-13; First posted 2015-09-15 (Estimated); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Tumors
Keywords: biliary; pancreatic; neuroendocrine; carcinoid; PNET; EP-NET; extrapancreatic; sarcoma; soft tissue sarcoma; STS; BTC
MeSH Terms: conditions — Neoplasms; Carcinoid Tumor; Neuroectodermal Tumors, Primitive; Sarcoma | interventions — surufatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Escalation 50 mg (Experimental): Escalation cohort at 50 mg/day
  Interventions: Drug: surufatinib
- Escalation 100mg (Experimental): Escalation cohort at 100 mg/day
  Interventions: Drug: surufatinib
- Escalation 200 mg (Experimental): Escalation cohort at 200 mg/day
  Interventions: Drug: surufatinib
- Escalation 300 mg (Experimental): Escalation cohort at 300 mg/day
  Interventions: Drug: surufatinib
- Escalation 400 mg (Experimental): Escalation cohort at 400 mg/day
  Interventions: Drug: surufatinib
- Expansion (Experimental): Subjects will receive RP2D surufatinib daily treatment continuously with every 28-day treatment cycle. Four expansion cohorts will enroll BTC, pNET, EP-NET, and STS patients, respectively.
  Interventions: Drug: surufatinib

INTERVENTIONS:
Drug: surufatinib — orally once daily (QD) in patients with advanced solid tumor.
  Other Names: HMPL-012; sulfatinib

SUMMARY:
Primary Objective Dose Escalation:

To evaluate the safety and tolerability of surufatinib in patients with advanced solid tumors and to determine the maximum tolerable dose (MTD) or recommended phase II dose (RP2D).

Primary Objective Dose Expansion:

To evaluate the anticancer activity of surufatinib in patients with advanced Biliary Tract Cancer (BTC), patients with advanced pancreatic neuroendocrine tumors (pNETs), patients with locally advanced, unresectable, metastatic extra-pancreatic neuroendocrine tumors (EP-NETs), and patients with soft tissue sarcomas (STS) treated at a dose of 300 mg QD.

Secondary Objective:

To evaluate the pharmacokinetic profile of multiple dose surufatinib in patients with advanced solid tumors and to evaluate the anti cancer activity of surufatinib in patients with advanced solid tumors.

DETAILED DESCRIPTION:
The study is an open-label, dose escalation and expansion clinical trial of surufatinib orally once daily (QD) in patients with advanced solid tumors.

The study consists of two phases:

Dose escalation phase - A 3+3 design will be used for this portion of the study.

* Approximately 15 to 35 evaluable patients will be enrolled. The actual number of patients depends on the Dose-limiting toxicity (DLT) situation as well as the RP2D dose level reached in this trial.
* The trial will approximately evaluate five surufatinib dose levels at 50,100, 200, 300 and 400 mg/day.

Expansion phase:

Approximately 115 patients will be enrolled into one of four open-label treatment arms during this phase: at least 30 patients with advanced BTC that has progressed on standard ﬁrst-line chemotherapy will be assigned to Arm A, at least 15 patients with advanced pNET that has progressed on either everolimus, sunitinib, or both will be assigned to Arm B, at least 15 patients with advanced EP-NET that has progressed on everolimus will be assigned to Arm C, and at least 45 patients with Soft Tissue Sarcoma will be assigned to Arm D. Subjects enrolled in this phase are to be evaluated for the safety, tolerability and pharmacokinetic (PK) characteristics to confirm the selected surufatinib dose.

Subjects will receive surufatinib daily treatment continuously with every 28-day treatment cycle until disease progression, death, or intolerable toxicity at the investigator's discretion for a favorable benefit to risk balance.

ELIGIBILITY:
Key Inclusion Criteria:

* Fully understand the study and voluntarily sign the informed consent form;
* At least 18 years old;
* Histologically or cytologically documented, locally advanced or metastatic solid malignancy of any type during the dose escalation phase, that has progressed on available standard systemic therapy, and for whom no effective therapy or standard of care exists; and locally advanced or metastatic BTC that has progressed on standard ﬁrst-line chemotherapy; locally advanced or metastatic pNET that has progressed on everolimus, sunitinib or both; locally advanced or metastatic EP-NET that has progressed on everolimus; advanced STS that has progressed on at least one line of standard therapy or refused standard frontline cytotoxic chemotherapy during the expansion phase;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Hypertension that is not controlled by antihypertension medication, defined as: systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg;
* History or presence of digestive tract diseases, including active gastric/duodenal ulcer or ulcerative colitis, or active hemorrhage of an unresected gastrointestinal tumor, or an evaluation by investigators of having any other condition that could possibly result in gastrointestinal tract hemorrhage or perforation;
* History or presence of serious hemorrhage , hemoptysis or hematemesis within 3 months or a thromboembolic event (including Deep Vein Thrombosis (DVT), stroke and/or transient ischemic attack) within 6 months;
* Patients with squamous Non Small Cell Lung Cancer (NSCLC) should be excluded;
* Clinically significant cardiovascular disease, including but not limited to, acute myocardial infarction within 6 months prior to enrollment, severe/unstable angina pectoris or coronary artery bypass grafting, New York Heart Association Class III/IV congestive heart failure, ventricular arrhythmias requiring treatment or left ventricular ejection fraction (LVEF) < 50%;
* Systemic anti-neoplastic therapies within 4 weeks prior to the initiation of investigational treatment, including chemotherapy, radical radiotherapy, hormonotherapy, biotherapy and immunotherapy;
* Palliative radiotherapy for bone metastasis/lesion within 2 weeks;
* Known Human immunodeficiency virus (HIV) infection;
* Known clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis;
* Women who are pregnant or lactating;
* Brain metastases and/or spinal cord compression untreated with surgery and/or radiotherapy, and without clinical imaging evidence of stable disease for 14 days or longer; Subjects requiring steroids within 4 weeks prior to start of study treatment will be excluded;
* Inability to take medication orally, dysphagia or an active gastric ulcer resulting from previous surgery or a severe gastrointestinal disease, or any other condition that investigators believe may affect absorption of the investigational product;
* Received investigational treatment in another clinical study within 4 weeks prior to the initiation of investigational treatment;
* Other disease, metabolic disorder, physical examination anomaly, abnormal laboratory result, or any other condition that investigators suspect may prohibit use of the investigational product, affect interpretation of study results, or put the patient at high risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marjo Hahka-Kemppinen, MD, PhD, Study Director — Hutchmed
Locations (12):
- United States (11):
  - City of Hope Comprehensive Cancer Center, Los Angeles, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - SCRI at HealthONE, Denver, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Tennessee Oncology, Nashville, Tennessee
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dasari A, Hamilton EP, Falchook GS, Wang JS, Li D, Sung MW, Chien C, Nanda S, Tucci C, Hahka-Kemppinen M, Paulson AS. A dose escalation/expansion study evaluating dose, safety, and efficacy of the novel tyrosine kinase inhibitor surufatinib, which inhibits VEGFR 1, 2, & 3, FGFR 1, and CSF1R, in US patients with neuroendocrine tumors. Invest New Drugs. 2023 Jun;41(3):421-430. doi: 10.1007/s10637-023-01359-2. Epub 2023 Apr 19. PMID 37074571

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 1/1b, 2-part, open-label study was conducted in patients with advanced solid tumors at 12 investigational sites in the United States and Italy.
Pre-assignment Details: The study consisted of a Dose-Escalation phase in patients with advanced solid tumors of any type and a Dose-Expansion phase in patients with advanced biliary tract cancer (BTC) (Arm A), advanced pancreatic neuroendocrine tumor (pNETs) (Arm B), advanced extrapancreatic neuroendocrine tumor (epNETs) (Arm C), or soft tissue sarcoma (STS) (Arm D). A total of 35 patients in Dose-Escalation phase and 95 patients in Dose-Expansion phase were enrolled in this study.
Groups:
- Dose-Escalation Phase: Surufatinib 50 Milligrams (mg): Patients received surufatinib 50 mg orally once daily (QD) throughout each 28-day treatment cycle until disease progression, death, intolerable toxicity, pregnancy, withdrawal of consent, or an Investigator's assessment that the patient can no longer benefit from the study drug.
- Dose-Escalation Phase: Surufatinib 100 mg: Patients received surufatinib 100 mg orally QD throughout each 28-day treatment cycle until disease progression, death, intolerable toxicity, pregnancy, withdrawal of consent, or an Investigator's assessment of loss of benefit from the study drug.
- Dose-Escalation Phase: Surufatinib 200 mg: Patients received surufatinib 200 mg orally QD throughout each 28-day treatment cycle until disease progression, death, intolerable toxicity, pregnancy, withdrawal of consent, or an Investigator's assessment of loss of benefit from the study drug.
- Dose-Escalation Phase: Surufatinib 300 mg: Patients received surufatinib 300 mg orally QD throughout each 28-day treatment cycle until disease progression, death, intolerable toxicity, pregnancy, withdrawal of consent, or an Investigator's assessment of loss of benefit from the study drug.
- Dose-Escalation Phase: Surufatinib 400 mg: Patients received surufatinib 400 mg orally QD throughout each 28-day treatment cycle until disease progression, death, intolerable toxicity, pregnancy, withdrawal of consent, or an Investigator's assessment of loss of benefit from the study drug.
- Dose-Expansion Phase: Arm A: BTC: Patients with advanced BTC received surufatinib 300 mg orally QD throughout each 28-day treatment cycle until disease progression, death, intolerable toxicity, pregnancy, withdrawal of consent, or an Investigator's assessment of loss of benefit from the study drug.
- Dose-Expansion Phase: Arm B: pNET: Patients with advanced pNET received surufatinib 300 mg orally QD throughout each 28-day treatment cycle until disease progression, death, intolerable toxicity, pregnancy, withdrawal of consent, or an Investigator's assessment of loss of benefit from the study drug.
- Dose-Expansion Phase: Arm C: epNET: Patients with advanced epNETs received surufatinib 300 mg orally QD throughout each 28-day treatment cycle until disease progression, death, intolerable toxicity, pregnancy, withdrawal of consent, or an Investigator's assessment of loss of benefit from the study drug.
- Dose-Expansion Phase: Arm D: STS: Patients with STS received surufatinib 300 mg orally QD throughout each 28-day treatment cycle until disease progression, death, intolerable toxicity, pregnancy, withdrawal of consent, or an Investigator's assessment of loss of benefit from the study drug.
Period: Overall Study
Arm/Group | Dose-Escalation Phase: Surufatinib 50 Milligrams (mg) | Dose-Escalation Phase: Surufatinib 100 mg | Dose-Escalation Phase: Surufatinib 200 mg | Dose-Escalation Phase: Surufatinib 300 mg | Dose-Escalation Phase: Surufatinib 400 mg | Dose-Expansion Phase: Arm A: BTC | Dose-Expansion Phase: Arm B: pNET | Dose-Expansion Phase: Arm C: epNET | Dose-Expansion Phase: Arm D: STS
Started | 3 | 7 | 3 | 9 | 13 | 30 | 16 | 16 | 33
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 7 | 3 | 9 | 13 | 30 | 16 | 16 | 33
Not completed — Death | 0 | 1 | 0 | 1 | 0 | 8 | 0 | 0 | 19
Not completed — No follow up required | 3 | 6 | 3 | 8 | 12 | 21 | 9 | 11 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 3 | 2
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Population: The Safety analysis set included all patients who received at least 1 dose of surufatinib.
Groups:
- Dose-Escalation Phase: Surufatinib 50 mg: Patients received surufatinib 50 mg orally QD throughout each 28-day treatment cycle until disease progression, death, intolerable toxicity, pregnancy, withdrawal of consent, or an Investigator's assessment that the patient can no longer benefit from the study drug.
- Total: Total of all reporting groups
Arm/Group | Dose-Escalation Phase: Surufatinib 50 mg | Dose-Escalation Phase: Surufatinib 100 mg | Dose-Escalation Phase: Surufatinib 200 mg | Dose-Escalation Phase: Surufatinib 300 mg | Dose-Escalation Phase: Surufatinib 400 mg | Dose-Expansion Phase: Arm A: BTC | Dose-Expansion Phase: Arm B: pNET | Dose-Expansion Phase: Arm C: epNET | Dose-Expansion Phase: Arm D: STS | Total
Number analyzed (Participants) | 3 | 7 | 3 | 9 | 13 | 30 | 16 | 16 | 33 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (4.16) | 58.1 (8.27) | 61.3 (7.04) | 62.6 (11.91) | 56.5 (13.20) | 65.6 (10.67) | 60.5 (10.72) | 61.4 (9.62) | 53.6 (13.48) | 59.4 (12.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 3 | 5 | 9 | 16 | 5 | 5 | 22 | 73
  Male | 1 | 1 | 0 | 4 | 4 | 14 | 11 | 11 | 11 | 57
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 4
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 6
  White | 2 | 7 | 3 | 9 | 12 | 29 | 6 | 9 | 26 | 103
  Other | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 2 | 6
  Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 2 | 10
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1 | 4 | 1 | 4 | 7 | 18
  Not Hispanic or Latino | 2 | 6 | 2 | 9 | 11 | 26 | 7 | 12 | 24 | 99
  Not Reported | 1 | 0 | 0 | 0 | 1 | 0 | 8 | 0 | 2 | 12
  Unknown | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Dose-Escalation Phase: Number of Patients With Dose-Limiting Toxicities (DLTs)
Description: A DLT was defined as any of the following toxicities determined by the Investigator to have a reasonable possibility of being related to surufatinib. Adverse events (AE) were graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Any Grade 4 non-hematological toxicity; any Grade 3 non-hematological toxicity except for nausea/vomiting, diarrhea, constipation, electrolyte imbalances, or transient hypertension downgraded within 3 days with appropriate supportive treatment; Grade 4 neutropenia lasting >7 days; Grade 3 febrile neutropenia (absolute neutrophil count <1.0 × 10^9/liter (L) with a single temperature of >38.3 degree Celsius (°C) or a sustained temperature of >=38°C for more than 1 hour; Grade 4 thrombocytopenia or >=Grade 3 thrombocytopenia associated with tendency to bleed; dose interruption or delay for >14 days due to toxicity; any life-threatening complication or abnormality not covered in NCI CTCAE v. 4.03.
Time Frame: From the first dose of study drug (Day 1) up to Day 28 of Cycle 1
Population: The DLT Evaluable set included all patients in Safety analysis set who were evaluable for DLT assessment. A patient was DLT evaluable if: had not received any preventive treatment during the DLT period and had completed the first 28-day treatment cycle with complete safety evaluations and had received at least 75% of the assigned surufatinib dose or had a confirmed DLT during the first 28-day treatment cycle.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-Escalation Phase: Surufatinib 50 mg | Dose-Escalation Phase: Surufatinib 100 mg | Dose-Escalation Phase: Surufatinib 200 mg | Dose-Escalation Phase: Surufatinib 300 mg | Dose-Escalation Phase: Surufatinib 400 mg
Number analyzed (Participants) | 3 | 6 | 3 | 9 | 11
Participants | 0 | 1 | 0 | 1 | 3

2. Primary Outcome: Dose-Escalation Phase: Number of Patients With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An AE was any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a drug or other protocol-imposed drug, regardless of attribution. An SAE was an AE that resulted in any of the following outcomes: was fatal; was life threatening; required or prolonged inpatient hospitalization; resulted in persistent or significant disability/incapacity; a congenital anomaly/birth defect in a neonate/infant born to a female patient or female partner of a male patient exposed to the study drug(s); was considered a significant medical event by the Investigator. TEAEs were defined as any AEs that started or worsened in severity on or after the first administration date of study drug and no later than 30 (+7) days after the last administration date of study drug or initiation of new anti-tumor therapy (whichever occurred first).
Time Frame: From the first dose of study drug (Day 1) up to approximately 90 months
Population: The Safety analysis set included all patients who received at least 1 dose of surufatinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-Escalation Phase: Surufatinib 50 mg | Dose-Escalation Phase: Surufatinib 100 mg | Dose-Escalation Phase: Surufatinib 200 mg | Dose-Escalation Phase: Surufatinib 300 mg | Dose-Escalation Phase: Surufatinib 400 mg
Number analyzed (Participants) | 3 | 7 | 3 | 9 | 13
Participants
  Any TEAEs | 3 | 7 | 3 | 9 | 13
  Any TESAEs | 1 | 2 | 0 | 4 | 4

3. Primary Outcome: Dose-Expansion Phase: Arms A and D: Progression Free Survival (PFS) Rate at 16 Weeks
Description: The tumor response was determined according to the international Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 guideline. PFS is defined as the time (in months) from the start date of study medication (Day 1) until the date of objective disease progression as defined by RECIST Version 1.1 or death (by any cause in the absence of progression), whichever occurred earlier. PFS rate probability at 16 week was estimated. Progression is defined by RECIST v1.0 as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (nadir), including baseline or appearance of 1 or more new lesions.
Time Frame: At 16 weeks
Population: The Safety analysis set included all patients who received at least 1 dose of surufatinib.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Dose-Expansion Phase: Arm A: BTC | Dose-Expansion Phase: Arm D: STS
Number analyzed (Participants) | 30 | 33
percentage of patients | 50.1 [27.8 to 68.9] | 26.5 [11.4 to 44.2]

4. Primary Outcome: Dose-Expansion Phase: Arms B and C: PFS Rate at 11 Months
Description: The tumor response was determined according to the RECIST v1.1 guideline. PFS is defined as the time (in months) from the start date of study medication (Day 1) until the date of objective disease progression as defined by RECIST Version 1.1 or death (by any cause in the absence of progression), whichever occurred earlier. PFS rate probability at 11 months was estimated. Progression is defined by RECIST v1.0 as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (nadir), including baseline or appearance of 1 or more new lesions.
Time Frame: At 11 months
Population: The Safety analysis set included all patients who received at least 1 dose of surufatinib.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Dose-Expansion Phase: Arm B: pNET | Dose-Expansion Phase: Arm C: epNET
Number analyzed (Participants) | 16 | 16
percentage of patients | 64.6 [34.7 to 83.5] | 60.9 [24.3 to 84.0]

5. Secondary Outcome: Dose-Escalation and Dose-Expansion Phase: Maximum Observed Plasma Concentration (Cmax) of Surufatinib
Description: Plasma samples were collected to determine Cmax of surufatinib. The pharmacokinetic (PK) parameters were determined by non-compartmental analysis.
Time Frame: Pre-dose and 1, 2, 4, 6, 8 hours post-dose on Days 1 and 15 of Cycle 1
Population: The PK analysis set included all patients whose plasma samples were collected for surufatinib concentration measurement and derivation of PK parameters. Combined data is presented for all patients evaluable for PK parameters who received surufatinib 300 mg in Dose-Escalation and Dose-Expansion phase. Only those patients with data collected at specified timepoints are reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Groups:
- Dose-Escalation and Dose-Expansion Phase: Surufatinib 300 mg: Patients received surufatinib 300 mg orally QD throughout each 28-day treatment cycle until disease progression, death, intolerable toxicity, pregnancy, withdrawal of consent, or an Investigator's assessment of loss of benefit from the study drug.
Arm/Group | Dose-Escalation Phase: Surufatinib 50 mg | Dose-Escalation Phase: Surufatinib 100 mg | Dose-Escalation Phase: Surufatinib 200 mg | Dose-Escalation and Dose-Expansion Phase: Surufatinib 300 mg | Dose-Escalation Phase: Surufatinib 400 mg
Number analyzed (Participants) | 3 | 7 | 3 | 79 | 13
nanogram/milliliter (ng/mL)
  Cycle 1 Day 1 | 73.6 (39.2) | 149 (107.3) | 180 (39.3) | 364 (66.6) | 427 (82.9)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 7 | 3 | 70 | 11
  Cycle 1 Day 15 | 99.0 (16.9) | 167 (109.0) | 261 (43.6) | 456 (68.0) | 566 (71.0)

6. Secondary Outcome: Dose Escalation and Dose-Expansion Phase: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Surufatinib
Description: Plasma samples were collected to determine Tmax of surufatinib. The PK parameters were determined by non-compartmental analysis.
Time Frame: Pre-dose and 1, 2, 4, 6, and 8 hours post-dose on Days 1 and 15 of Cycle 1
Population: as for outcome 5
Measure: Median (Full Range); unit: hour
Arm/Group | Dose-Escalation Phase: Surufatinib 50 mg | Dose-Escalation Phase: Surufatinib 100 mg | Dose-Escalation Phase: Surufatinib 200 mg | Dose-Escalation and Dose-Expansion Phase: Surufatinib 300 mg | Dose-Escalation Phase: Surufatinib 400 mg
Number analyzed (Participants) | 3 | 7 | 3 | 79 | 13
hour
  Cycle 1 Day 1 | 2.00 [1.02 to 2.17] | 1.03 [1.00 to 4.00] | 2.05 [1.02 to 3.58] | 2.20 [0.75 to 23.7] | 3.83 [1.18 to 8.13]
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 7 | 3 | 70 | 11
  Cycle 1 Day 15 | 3.98 [1.97 to 4.00] | 2.00 [0.98 to 3.88] | 2.03 [1.00 to 2.12] | 3.50 [0.73 to 7.88] | 4.00 [2.00 to 7.07]

7. Secondary Outcome: Dose-Escalation and Dose-Expansion Phase: Area Under the Plasma Concentration-Time Curve From Time 0 to 24 Hours (AUC0-24h) of Surufatinib
Description: Plasma samples were collected to determine AUC0-24h of surufatinib. The PK parameters were determined by non-compartmental analysis. Data from pre-dose to 8 hours post-dose were extrapolated to obtain the AUC0-24 data.
Time Frame: Pre-dose and 1, 2, 4, 6, and 8 hours post-dose on Cycle 1 Day 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | Dose-Escalation Phase: Surufatinib 50 mg | Dose-Escalation Phase: Surufatinib 100 mg | Dose-Escalation Phase: Surufatinib 200 mg | Dose-Escalation and Dose-Expansion Phase: Surufatinib 300 mg | Dose-Escalation Phase: Surufatinib 400 mg
Number analyzed (Participants) | 3 | 7 | 3 | 68 | 12
hour*ng/mL | 616 (7.5) | 877 (81.2) | 1360 (10.5) | 3080 (58.8) | 3540 (76.8)

8. Secondary Outcome: Dose-Escalation and Dose-Expansion Phase: AUC Over the Dosing Interval (AUCtau) of Surufatinib
Description: Plasma samples were collected to determine AUCtau of surufatinib. The PK parameters were determined by non-compartmental analysis.
Time Frame: Pre-dose and 1, 2, 4, 6, and 8 hours post-dose on Day 15 of Cycle 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | Dose-Escalation Phase: Surufatinib 50 mg | Dose-Escalation Phase: Surufatinib 100 mg | Dose-Escalation Phase: Surufatinib 200 mg | Dose-Escalation and Dose-Expansion Phase: Surufatinib 300 mg | Dose-Escalation Phase: Surufatinib 400 mg
Number analyzed (Participants) | 3 | 7 | 3 | 67 | 10
hour*ng/mL | 968 (1.5) | 1320 (95.2) | 2310 (36.7) | 4770 (64.4) | 6890 (60.5)

9. Secondary Outcome: Dose-Escalation and Dose-Expansion Phase: Objective Response Rate (ORR)
Description: The ORR was defined as the percentage of patients achieving a complete response (CR) or partial response (PR) as confirmed best overall response (BOR) as determined by the Investigator using RECIST v1.1. The BOR was defined as the best response recorded from the start of study treatment until documented RECIST version 1.1 progression, death, or withdrawal of consent. The CR was defined as disappearance of all target lesions. The PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: RECIST assessments performed at screening (within 28 days before start of study treatment), Day 1 of Cycle 2, and every 8 (+/-1 week) weeks afterwards until the occurrence of disease progression, up to a maximum of 90 months
Population: The Efficacy analysis set included all patients who received at least 1 dose of surufatinib and had at least 1 post-baseline tumor assessment.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Dose-Escalation Phase: Surufatinib 50 mg | Dose-Escalation Phase: Surufatinib 100 mg | Dose-Escalation Phase: Surufatinib 200 mg | Dose-Escalation Phase: Surufatinib 300 mg | Dose-Escalation Phase: Surufatinib 400 mg | Dose-Expansion Phase: Arm A: BTC | Dose-Expansion Phase: Arm B: pNET | Dose-Expansion Phase: Arm C: epNET | Dose-Expansion Phase: Arm D: STS
Number analyzed (Participants) | 3 | 6 | 3 | 8 | 11 | 27 | 16 | 16 | 30
percentage of patients | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 36.9] | 9.1 [0.2 to 41.3] | 0.0 [0.0 to 12.8] | 18.8 [4.0 to 45.6] | 6.3 [0.2 to 30.2] | 0.0 [0.0 to 11.6]

10. Secondary Outcome: Dose-Escalation and Dose-Expansion Phase: Disease Control Rate (DCR)
Description: The DCR was defined as the percentage of patients who achieved a CR, PR or stable disease (SD) as confirmed BOR as determined by the Investigator using RECIST v1.1. The CR was defined as disappearance of all target lesions. The PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum on study.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Dose-Escalation Phase: Surufatinib 50 mg | Dose-Escalation Phase: Surufatinib 100 mg | Dose-Escalation Phase: Surufatinib 200 mg | Dose-Escalation Phase: Surufatinib 300 mg | Dose-Escalation Phase: Surufatinib 400 mg | Dose-Expansion Phase: Arm A: BTC | Dose-Expansion Phase: Arm B: pNET | Dose-Expansion Phase: Arm C: epNET | Dose-Expansion Phase: Arm D: STS
Number analyzed (Participants) | 3 | 6 | 3 | 8 | 11 | 27 | 16 | 16 | 30
percentage of patients | 33.3 [0.8 to 90.6] | 50.0 [11.8 to 88.2] | 33.3 [0.8 to 90.6] | 50.0 [15.7 to 84.3] | 72.7 [39.0 to 94.0] | 48.1 [28.7 to 68.1] | 87.5 [61.7 to 98.4] | 93.8 [69.8 to 99.8] | 30.0 [14.7 to 49.4]

11. Secondary Outcome: Dose-Escalation and Dose-Expansion Phase: Duration of Response (DoR)
Description: The DoR was defined as the time from the first time that the objective response reached CR or PR, whichever came first (and later confirmed), until the occurrence of PD or death. The CR was defined as disappearance of all target lesions. The PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. The PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (nadir), including baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters. The appearance of 1 or more new lesions was also considered progression.
Time Frame: as for outcome 9
Population: The Efficacy analysis set included all patients who received at least 1 dose of surufatinib and had at least 1 post-baseline tumor assessment. Only those patients with PR or CR (responders) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose-Escalation Phase: Surufatinib 50 mg | Dose-Escalation Phase: Surufatinib 100 mg | Dose-Escalation Phase: Surufatinib 200 mg | Dose-Escalation Phase: Surufatinib 300 mg | Dose-Escalation Phase: Surufatinib 400 mg | Dose-Expansion Phase: Arm A: BTC | Dose-Expansion Phase: Arm B: pNET | Dose-Expansion Phase: Arm C: epNET | Dose-Expansion Phase: Arm D: STS
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 0
months |  |  |  |  | 13.142 [NA to NA] — NA indicates that upper and lower limits of confidence interval (CI) were not estimable due to insufficient number of patients with events at study closure. |  | NA [14.752 to NA] — NA indicates that median and upper limit of CI were not estimable due to insufficient number of patients with events at study closure. | 14.784 [NA to NA] — NA indicates that upper and lower limits of CI were not estimable due to insufficient number of patients with events at study closure. |

12. Secondary Outcome: Dose-Escalation Phase: Progression-Free Survival (PFS)
Description: The PFS was defined as the time from the start date of study drug until the date of objective PD as assessed by the Investigator using RECIST version 1.1 or death (by any cause in the absence of progression).
Time Frame: RECIST assessments performed at screening (within 28 days before start of study treatment), Day 1 of Cycle 2, and every 8 (+/-1 week) weeks afterwards until the occurrence of disease progression, up to a maximum of 53 months
Population: The Safety analysis set included all patients who received at least 1 dose of surufatinib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose-Escalation Phase: Surufatinib 50 mg | Dose-Escalation Phase: Surufatinib 100 mg | Dose-Escalation Phase: Surufatinib 200 mg | Dose-Escalation Phase: Surufatinib 300 mg | Dose-Escalation Phase: Surufatinib 400 mg
Number analyzed (Participants) | 3 | 7 | 3 | 9 | 13
months | 2.793 [1.873 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure. | 2.530 [0.887 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure. | 5.322 [0.920 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure. | 2.694 [1.676 to 3.680] | 8.378 [1.741 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure.

13. Secondary Outcome: Dose-Expansion Phase: Time to Response (TTR)
Description: The TTR was defined as the time from the start of study drug until first documented response (and later confirmed) according to RECIST v.1.1 for responders only.
Time Frame: as for outcome 12
Population: The Efficacy analysis set included all patients who received at least 1 dose of study medication and had at least 1 post-baseline tumor assessment. Only those patients who achieved CR/PR (responders) were included in the analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Dose-Expansion Phase: Arm A: BTC | Dose-Expansion Phase: Arm B: pNET | Dose-Expansion Phase: Arm C: epNET | Dose-Expansion Phase: Arm D: STS
Number analyzed (Participants) | 0 | 3 | 1 | 0
months |  | 2.760 [2.69 to 4.63] | 2.497 [2.497 to 2.497] |

14. Secondary Outcome: Dose-Escalation and Dose-Expansion Phase: Maximum Percentage Change From Baseline in Tumor Size as Per RECIST v1.1
Description: Percentage change in tumor size was determined for patients with measurable disease at baseline and was derived at each visit by the percentage change in the sum of the diameters of target lesions compared to baseline, mean of maximum percentage change is presented. Baseline was defined as the last evaluable tumor assessment result obtained prior to the administration of study drug (including unscheduled assessments).
Time Frame: as for outcome 9
Population: The Efficacy analysis set included all patients who received at least 1 dose of surufatinib and had at least 1 post-baseline tumor assessment. Only those patients with data collected are reported.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Dose-Escalation Phase: Surufatinib 50 mg | Dose-Escalation Phase: Surufatinib 100 mg | Dose-Escalation Phase: Surufatinib 200 mg | Dose-Escalation Phase: Surufatinib 300 mg | Dose-Escalation Phase: Surufatinib 400 mg | Dose-Expansion Phase: Arm A: BTC | Dose-Expansion Phase: Arm B: pNET | Dose-Expansion Phase: Arm C: epNET | Dose-Expansion Phase: Arm D: STS
Number analyzed (Participants) | 1 | 6 | 3 | 8 | 11 | 25 | 16 | 16 | 30
percentage change | -17.895 (NA) — NA indicates that standard deviation cannot be derived for a single patient. | -14.076 (42.9290) | 2.925 (19.8263) | 7.982 (21.9026) | -10.249 (38.9841) | -2.129 (19.5407) | -15.210 (28.1133) | -11.047 (12.8727) | 6.658 (25.1689)

ADVERSE EVENTS:
Time Frame: TEAEs and all-cause mortality were collected from the first dose of study drug (Day 1) up to approximately 90 months
Description: The Safety analysis set included all patients who received at least 1 dose of surufatinib.
Arm/Group | Dose-Escalation Phase: Surufatinib 50 mg | Dose-Escalation Phase: Surufatinib 100 mg | Dose-Escalation Phase: Surufatinib 200 mg | Dose-Escalation Phase: Surufatinib 300 mg | Dose-Escalation Phase: Surufatinib 400 mg | Dose-Expansion Phase: Arm A: BTC | Dose-Expansion Phase: Arm B: pNET | Dose-Expansion Phase: Arm C: epNET | Dose-Expansion Phase: Arm D: STS
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/7 | 0/3 | 1/9 | 0/13 | 8/30 | 0/16 | 0/16 | 20/33
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/7 | 0/3 | 4/9 | 4/13 | 11/30 | 8/16 | 7/16 | 15/33
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 3/3 | 9/9 | 13/13 | 26/30 | 15/16 | 16/16 | 31/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose-Escalation Phase: Surufatinib 50 mg (N=3) | Dose-Escalation Phase: Surufatinib 100 mg (N=7) | Dose-Escalation Phase: Surufatinib 200 mg (N=3) | Dose-Escalation Phase: Surufatinib 300 mg (N=9) | Dose-Escalation Phase: Surufatinib 400 mg (N=13) | Dose-Expansion Phase: Arm A: BTC (N=30) | Dose-Expansion Phase: Arm B: pNET (N=16) | Dose-Expansion Phase: Arm C: epNET (N=16) | Dose-Expansion Phase: Arm D: STS (N=33)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epiglottitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose-Escalation Phase: Surufatinib 50 mg (N=3) | Dose-Escalation Phase: Surufatinib 100 mg (N=7) | Dose-Escalation Phase: Surufatinib 200 mg (N=3) | Dose-Escalation Phase: Surufatinib 300 mg (N=9) | Dose-Escalation Phase: Surufatinib 400 mg (N=13) | Dose-Expansion Phase: Arm A: BTC (N=30) | Dose-Expansion Phase: Arm B: pNET (N=16) | Dose-Expansion Phase: Arm C: epNET (N=16) | Dose-Expansion Phase: Arm D: STS (N=33)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (5) | 1 (1) | 4 (5) | 7 (9) | 8 (8) | 5 (6) | 5 (9) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 3 (5) | 0 (0) | 2 (3) | 10 (18) | 11 (18) | 7 (10) | 6 (11) | 9 (15)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 4 (5) | 7 (8) | 4 (6) | 5 (6) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 4 (4) | 7 (11) | 6 (7) | 3 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 2 (2) | 5 (6) | 4 (4) | 4 (4) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 5 (5) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (4) | 2 (2)
Fatigue (General disorders) | 1 (1) | 4 (8) | 0 (0) | 2 (4) | 6 (9) | 8 (13) | 5 (11) | 10 (14) | 13 (16)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 6 (7) | 6 (6) | 1 (1) | 6 (6)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (5) | 3 (4) | 2 (4) | 1 (4)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 2 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 5 (5) | 4 (5) | 5 (5) | 3 (3)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 4 (6) | 2 (2) | 3 (7)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 2 (2) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 5 (6) | 3 (3) | 5 (6) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (3) | 3 (3) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 1 (2) | 3 (3) | 6 (6)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 4 (4) | 6 (7) | 4 (5) | 5 (8)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 2 (4) | 5 (5)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 4 (7) | 13 (17) | 8 (10) | 7 (10) | 12 (15)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (11) | 8 (21) | 8 (22) | 7 (15) | 7 (7)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (4) | 2 (2) | 3 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 3 (5) | 2 (4) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 3 (6) | 1 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 5 (15) | 3 (3) | 1 (1) | 6 (8)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 3 (3) | 2 (4) | 2 (3) | 1 (2)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (4) | 4 (5) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 3 (4) | 4 (4) | 3 (3)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (5) | 1 (2) | 2 (3) | 4 (4)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 3 (3) | 3 (6) | 3 (5) | 4 (7)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 5 (6) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT02549937/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT02549937/SAP_001.pdf